CLINICAL TRIAL: NCT00365352
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of XP13512 in Patients With Restless Legs Syndrome.
Brief Title: XP13512 vs. Placebo in Patients With Restless Legs Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111460; XP053 (Other: XenoPort, Inc.)
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- XP13512 600MG (Experimental): XP13512 600MG ONCE DAILY
  Interventions: Drug: XP13512 600MG
- XP13512 1200MG (Experimental): XP13512 1200MG ONCE DAILY
  Interventions: Drug: XP13512 1200MG
- Placebo (Placebo Comparator): PLACEBO ONCE DAILY
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: XP13512 600MG — XP13512 600MG ONCE DAILY
  Other Names: GSK1838262; Gabapentin Enacarbil
  Arms: XP13512 600MG
Drug: XP13512 1200MG — XP13512 1200MG ONCE DAILY
  Other Names: GSK1838262; Gabapentin Enacarbil
  Arms: XP13512 1200MG
Drug: PLACEBO — PLACEBO ONCE DAILY
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the efficacy of XP13512 taken once daily compared to placebo for the treatment of patients suffering from Restless Legs Syndrome (RLS).

DETAILED DESCRIPTION:
This was a 12-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the efficacy and safety of XP13512 in subjects with Restless Legs Syndrome (RLS). Eligible subjects were randomized to receive 1 of 3 once daily oral doses of XP13512 1200 mg, XP13512 600 mg, or placebo. The primary study objective was to compare the efficacy of XP13512 1200 mg taken once daily for 12 weeks versus placebo. The secondary study objectives were to assess the efficacy of XP13512 600 mg taken once daily for the reatment of RLS and to assess the onset of treatment benefits and improvement in sleep, pain, mood, quality of life, and safety and tolerability of both XP13512 1200 mg and 600 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary RLS, based on the International RLS Study Diagnostic Criteria.

Exclusion Criteria:

* A sleep disorder (e.g., sleep apnea) that may significantly affect the assessment of RLS;
* Neurologic disease or movement disorder (e.g., diabetic neuropathy, Parkinson's Disease, Multiple Sclerosis, dyskinesias, and dystonias);
* Abnormal laboratory results, electrocardiogram (ECG) or physical findings;
* Pregnant or lactating women;
* Women of childbearing potential who are not practicing an acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Ahmed M, Hays R, Steven Poceta J, Jaros MJ, Kim R, Shang G. Effect of Gabapentin Enacarbil on Individual Items of the International Restless Legs Study Group Rating Scale and Post-sleep Questionnaire in Adults with Moderate-to-Severe Primary Restless Legs Syndrome: Pooled Analysis of 3 Randomized Trials. Clin Ther. 2016 Jul;38(7):1726-1737.e1. doi: 10.1016/j.clinthera.2016.05.008. Epub 2016 Jun 7. PMID 27288210
- [Derived] Avidan AY, Lee D, Park M, Jaros MJ, Shang G, Kim R. The Effect of Gabapentin Enacarbil on Quality of Life and Mood Outcomes in a Pooled Population of Adult Patients with Moderate-to-Severe Primary Restless Legs Syndrome. CNS Drugs. 2016 Apr;30(4):305-16. doi: 10.1007/s40263-016-0329-4. PMID 27067343
- [Derived] Ondo WG, Hermanowicz N, Borreguero DG, Jaros MJ, Kim R, Shang G. Effect of prior exposure to dopamine agonists on treatment with gabapentin enacarbil in adults with moderate-to-severe primary restless legs syndrome: pooled analyses from 3 randomized trials. J Clin Mov Disord. 2015 Mar 30;2:9. doi: 10.1186/s40734-015-0018-3. eCollection 2015. PMID 26788345
- [Derived] Lee DO, Ziman RB, Perkins AT, Poceta JS, Walters AS, Barrett RW; XP053 Study Group. A randomized, double-blind, placebo-controlled study to assess the efficacy and tolerability of gabapentin enacarbil in subjects with restless legs syndrome. J Clin Sleep Med. 2011 Jun 15;7(3):282-92. doi: 10.5664/JCSM.1074. PMID 21677899
- [Derived] Canafax DM, Bhanegaonkar A, Bharmal M, Calloway M. Validation of the post sleep questionnaire for assessing subjects with restless legs syndrome: results from two double-blind, multicenter, placebo-controlled clinical trials. BMC Neurol. 2011 Apr 28;11:48. doi: 10.1186/1471-2377-11-48. PMID 21527006

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral placebo tablet taken once daily. Days 1 to 3: one placebo tablet. Days 4 to 84: two placebo tablets. On Days 85 participants entered a 7-day Taper Period. Days 85 to 91: one placebo tablet.
- GEn (XP13512/GSK1838262) 600 mg: Gabapentin enacarbil (GEn) (XP13512/GSK1838262) 600 milligrams (mg) taken orally once a day for 12 weeks) taken once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 84: one ER tablet (600 mg GEn) and one placebo tablet. On Day 85, participants entered a 7-day Taper Period. Days 85 to 91: one placebo tablet.
- GEn (XP13512/GSK1838262) 1200 mg: Oral GEn (gabapentin enacarbil) 1200 milligrams (mg) taken once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 84: two ER tablets (1200 mg GEn). On Day 85, participants entered a 7-day Taper Period. Days 85 to 91: one ER tablet (600 mg GEn).
Period: Overall Study
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Started | 97 | 115 | 113
Safety Population | 96 | 115 | 111
Modified Intent-to-Treat Population | 96 | 114 | 111
Completed | 77 | 104 | 98
Not Completed | 20 | 11 | 15
Not completed — Adverse Event | 6 | 7 | 8
Not completed — Participant Withdrew Consent | 8 | 3 | 4
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Ineligible (Did Not Meet Entry Criteria) | 0 | 0 | 2
Not completed — Non-Compliance (after Randomization) | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal of Participant by Sponsor | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg | Total
Number analyzed (Participants) | 96 | 114 | 111 | 321
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were collected from members of the Modified Intent-to-Treat (MITT) Population, comprised of all participants in the Safety Population who also satisfied both of the following conditions: (1) completed the International Restless Legs Syndrome (IRLS) Rating Scale at Baseline; and (2) completed at least one on-treatment IRLS Rating Scale score during the treatment period.
  Years | 49.1 (12.19) | 48.3 (12.88) | 49.5 (12.67) | 48.9 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristics were collected for members of the Modified Intent-to-Treat (MITT) Population, comprised of all participants in the Safety Population who also satisfied both of the following conditions: (1) completed the International Restless Legs Syndrome (IRLS) Rating Scale at Baseline; and (2) completed at least one on-treatment IRLS Rating Scale score during the treatment period.
  Participants
    Female | 57 | 66 | 65 | 188
    Male | 39 | 48 | 46 | 133
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristics were collected in members of the Modified Intent-to-Treat (MITT) Population, comprised of all participants in the Safety Population who also satisfied both of the following conditions: (1) completed the International Restless Legs Syndrome (IRLS) Rating Scale at Baseline; and (2) completed at least one on-treatment IRLS Rating Scale score during the treatment period. Patients were allowed to categorize to more than one race.
  participants
    American Indian or Alaskan Native | 1 | 3 | 0 | 4
    Asian | 2 | 0 | 1 | 3
    Black or African American | 1 | 5 | 1 | 7
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    White or Caucasian | 92 | 106 | 107 | 305
    Unknown | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in IRLS Rating Scale Total Score at Week 12 Using Last Observation Carried Forward (LOCF)
Description: The International Restless Legs Syndrome (IRLS) Rating scale is a measure of RLS disease severity. The scale reflects the participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Ten items (individually scored from 0 to 4) are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total scale score is a sum of all of the individual item scores and ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement.
Time Frame: Baseline and Week 12
Population: Modified Intent-to-Treat (MITT) Population: all participants in the Safety Population who also satisfied all of the following conditions: (1) completed the IRLS Rating Scale at Baseline; and (2) completed at least one on-treatment IRLS Rating Scale score during the treatment period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 111
scores on a scale | -9.8 (7.69) | -13.0 (9.12)
Statistical Analysis 1: Comparison: Placebo vs GEn (XP13512/GSK1838262) 1200 mg; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Final Values) = -3.5, 95% CI [-5.6 to -1.3] — Mean difference was adjusted for Baseline value, treatment pooled sites, and treatment by pool site interaction

2. Primary Outcome: Number of Participants With a Score of "Much Improved" or "Very Much Improved" on the Investigator-rated CGI-I Scale (Response) at (Week 12) Using LOCF
Description: The investigator -rated Clinical Global Impression of Improvement (CGI-I) scale is an assessment designed to allow investigators to rate the change of a participant's disease severity over time based on a seven-point scale, with a score of 1 being "very much improved," a score of 2 being "much improved," a score of 3 being "minimally improved," a score of 4 being "no change," a score of 5 being "minimally improved,"a score of 6 being "much worse," and a score of 7 being "very much worse." Participants with a response of "much improved" or "very much improved" were classified as responders.
Time Frame: Week 12
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 111
participants | 43 | 86
Statistical Analysis 1: Comparison: Placebo vs GEn (XP13512/GSK1838262) 1200 mg; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; A logistic regression model was used with treatment and pooled center as explanatory factors; Odds Ratio (OR) = 4.287, 95% CI [2.338 to 7.861]

3. Secondary Outcome: Change From Baseline to the End of Treatment (Week 12) in the IRLS Rating Scale Total Score Using LOCF
Description: The IRLS Rating scale is a measure of RLS disease severity. The scale reflects the participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Items (individually scored from 0 to 4) are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total scale score is a sum of all of the individual item scores and ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement.
Time Frame: Baseline (Day 1) and End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg
Number analyzed (Participants) | 96 | 114
scores on a scale | -9.8 (7.69) | -13.8 (8.09)

4. Secondary Outcome: Number of Participants Classsified as Responders on the Investigator-rated CGI-I Scale at Week 12 Using LOCF
Description: The CGI-I scale is a standardized tool that is widely used in psychopharmacologic trials. For the CGI-I, the investigator was asked to rate the participant's overall change in RLS symptoms from Baseline. Scores ranged from 1 (very much improved) to 7 (very much worse). Participants who were much improved (score of 2) or very much improved on the CGI-I scale at the end of treatment (Week 12) are classified as "Responders."
Time Frame: Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg
Number analyzed (Participants) | 96 | 114
participants | 43 | 83

5. Secondary Outcome: Number of Participants Who Had an Onset of Response to Treatment at the End of Week 1 Based Upon the IRLS Rating Scale Total Score and the Investigator-rated CGI-I Using LOCF
Description: The IRLS Rating scale is a measure of RLS disease severity. Items (individually scored from 0 to 4) are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total scale score is a sum of all of the individual item scores and ranges from 0-40 points, with 40 being the most severe. Response was defined by an IRLS Rating Scale total score at the end of Week 1 < 15 and at least a 6-point reduction from the participant's Baseline score and an investigator-rated CGI-I response of "much improved" or "very much improved."
Time Frame: End of Week 1
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
participants | 13 | 36 | 40

6. Secondary Outcome: The Time to Onset of the First Response to Treatment on the IRLS Rating Scale Total Score and the Investigator-rated CGI-I
Description: The Response was defined by an IRLS Rating Scale total score at the end of Week 1 < 15 and at least a 6-point reduction from the participant's Baseline score and an investigator-rated CGI-I response of much improved or very much improved. The median time to onset is estimated using the product-limit estimation method.
Time Frame: Baseline (Day 1) to End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- GEn (XP13512/GSK1838262) 600 Milligrams(mg) Taken Orally: Gabapentin enacarbil (GEn) (XP13512/GSK1838262) 600 milligrams (mg) taken orally once a day for 12 weeks) taken once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 84: one ER tablet (600 mg GEn) and one placebo tablet. On Day 85, participants entered a 7-day Taper Period. Days 85 to 91: one placebo tablet.
- GEn (XP13512/GSK1838262) 1200 mg Taken Orally Once a Day: Oral GEn (gabapentin enacarbil) 1200 milligrams (mg) taken once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 84: two ER tablets (1200 mg GEn). On Day 85, participants entered a 7-day Taper Period. Days 85 to 91: one ER tablet (600 mg GEn).
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 Milligrams(mg) Taken Orally | GEn (XP13512/GSK1838262) 1200 mg Taken Orally Once a Day
Number analyzed (Participants) | 96 | 114 | 111
weeks | NA [NA to NA] — The median value was not estimable because fewer than 50% of the participants experienced the event. | 4.1 [2.1 to 8.1] | 2.1 [2.1 to 4.0]

7. Secondary Outcome: Mean Change in the IRLS Rating Scale Total Score From Baseline at Week 12 by RLS Treatment History Using LOCF
Description: The IRLS Rating scale is a measure of RLS disease severity. The scale reflects the participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Ten items (individually scored from 0 to 4) are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total scale score is a sum of all of the individual item scores and ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement.
Time Frame: Baseline (Day 1) and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale
  No RLS Treatment History | -8.8 (7.08) | -13.7 (8.23) | -12.5 (8.78)
  Treatment terminated | -13.3 (9.09) | -12.4 (7.26) | -17.1 (7.94)
  Treatment within 1 month of study start | -10.7 (8.11) | -14.6 (8.39) | -12.1 (10.43)

8. Secondary Outcome: Change From Baseline in the IRLS Rating Scale Total Score at Week 12 by Baseline RLS Rating Scale Total Score Category (Baseline RLS Severity) Using LOCF
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale
  IRLS Total Score < 17.5 | -6.3 (4.98) | -8.9 (6.02) | -7.9 (6.81)
  IRLS Total Score 17.5 to < 22.5 | -8.5 (7.11) | -11.9 (6.34) | -8.8 (7.77)
  IRLS Total Score 22.5 to < 27.5 | -9.6 (8.21) | -15.1 (6.65) | -15.5 (8.12)
  IRLS Total Score >= 27.5 | -13.3 (7.74) | -18.2 (11.28) | -19.6 (8.80)

9. Secondary Outcome: Change From Baseline to the End of Week 1 in the IRLS Rating Scale Total Score Using LOCF
Description: as for outcome 3
Time Frame: Baseline and the End of Week 1
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale | -6.0 (5.59) | -9.8 (7.76) | -8.7 (8.09)

10. Secondary Outcome: Number of Participants Classified as Investigator-rated CGI-I Scale Responders at Week 12 by RLS Treatment History Using LOCF
Description: as for outcome 4
Time Frame: Basline and Week 12
Population: Participants included in the MITT Population with a known RLS treatment history
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 94 | 112 | 110
participants
  No RLS Treatment History | 26 | 54 | 57
  Treatment terminated | 5 | 9 | 13
  Treatment within 1 month of study start | 11 | 18 | 15

11. Secondary Outcome: Number of Total Responders to Treatment Based on the Investigator-Rated CGI of Improvement at the End of One Week of Treatment
Description: as for outcome 4
Time Frame: End of Week 1
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: responders
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
responders | 26 | 54 | 59

12. Secondary Outcome: Change From Baseline to the End of Treatment in Average Daily Total Sleep Time (Hours) Using LOCF
Description: Average daily total sleep time was derived from the Pittsburgh Sleep Diary (PghSD; an instrument with separate components to be completed [self-reported] at bedtime and waketime) as the mean of non-missing total sleep time over the 7 days before each visit, where total sleep time = [(wake up time - lights out time) - time to fall asleep - time awake during the night] in hours. The change was calculated as the end of treatment (Week 12) value minus the Baseline value.
Time Frame: Baseline to End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 113 | 111
hours | 0.6 (1.36) | 0.7 (1.25) | 1.0 (1.32)

13. Secondary Outcome: Change From Baseline to the End of Treatment in Average Daily Wake Time (Minutes) After Sleep Onset Using LOCF
Description: Average daily wake time after sleep onset was derived from the Pittsburgh Sleep Diary (PghSD) as the mean of non-missing total hours awake during the night after falling asleep over the 7 days before each visit. The change was calculated as the end of treatment (Week 12) value minus the Baseline value.
Time Frame: Baseline to End of Treatment (Week 12)
Population: MITT Popultion. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 113 | 111
minutes | -12.5 (31.01) | -16.4 (22.33) | -18.5 (28.67)

14. Secondary Outcome: Change From Baseline in the Average Daily RLS Pain Score at the End of Treatment (Week 12) for Participants With Pain at Baseline or the End of Week 12 Using LOCF
Description: The Daily RLS pain score was assessed by participants reporting whether they experienced any pain associated with RLS in the last 24 hours and rating their pain levels on an 11-point numerical rating scale, with 0 being no pain and 10 the most intense pain imaginable. The assessment was performed for 7 days prior to Baseline and pre-defined study visits. The change from baseline was calculated as the End of Treatment (Week 12) value minus the Baseline (Day 1) value.
Time Frame: Baseline and End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale | -1.7 (2.28) | -2.5 (2.20) | -2.6 (2.43)

15. Secondary Outcome: Number of Participants Classified as Responders With at Least 30% and 50% Improvement in the Average Daily RLS Pain Score Using LOCF
Description: The Mean Daily RLS pain was assessed by participants reporting whether they experienced any pain associated with RLS in the last 24 hours and rating their pain levels on an 11-point numerical rating scale, with 0 being no pain and 10 the most intense pain imaginable. The assessment was performed for 7 days prior to Baseline and pre-defined visits A "Responder" is a participant with a score of "much improved" or "very much improved" on the investigator rated CGI I Scale at the end of treatment (Week 12 using LOCF).
Time Frame: Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
participants
  > or equal to 30% response | 48 | 75 | 76
  > or equal to 50% response | 41 | 62 | 66

16. Secondary Outcome: Change From Baseline in the Average Daily RLS Pain Score to Week 12 for Participants With a Baseline Pain Score of at Least 4 Using LOCF
Description: The Average Daily RLS pain was assessed by participants reporting whether they experienced any pain associated with RLS in the last 24 hours and rating their pain levels on an 11-point numerical rating scale, with 0 being no pain and 10 the most intense pain imaginable. The assessment was performed for 7 days prior to Baseline and pre-defined visits. The change from baseline was calculated as the End of Treatment (Week 12) value minus the Baseline (Day 1) value.
Time Frame: Baseline and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale | -2.3 (2.34) | -3.5 (2.19) | -3.5 (2.51)

17. Secondary Outcome: Number of Participants Classified as Responders to Treatment Based on the Participant-Rated CGI of Improvement at Week 1 and Week 12 (End of Treatment)
Description: as for outcome 4
Time Frame: Week 1 and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
participants
  Responders at the End of Treatment (Week 12) | 46 | 90 | 83
  Responders at the End of One Week | 20 | 55 | 52

18. Secondary Outcome: Number of Participants With a Rating of Excellent for the Overall Quality of Sleep in Past Week Measured by the Post-Sleep Questionnaire (PSQ) at the End of Treatment (Week 12) Using LOCF
Description: The Post-Sleep Questionnaire (PSQ) was designed to evaluate overall sleep quality, ability to function, and RLS symptoms' interference with sleep over the past week. Participants were asked to rate overall sleep quality (as either "Excellent," "Reasonable," or "Poor"), ability to function, number of nights with RLS symptoms, number of nights awakened by RLS symptoms, and the number of hours spent awake due to RLS symptoms over the past week.
Time Frame: End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
participants | 14 | 24 | 30

19. Secondary Outcome: Number of Participants Who Indicated on the Mood Assessment That Their Mood Was Much Improved or Very Much Improved at Week 12 (End of Treatment) Using LOCF
Description: The Mood Assessment is a non-disease-specific question surveying global change in a participant's overall mood. Participants were asked to rate their overall change in mood since the start of the study by choosing a score in a range from 1 (Very Much Improved) to 7 (Very Much Worse). The assessment was completed at Day 1 and the ends of Weeks 4, 8, and 12 or (Early Termination).
Time Frame: Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
participants | 19 | 35 | 39

20. Secondary Outcome: Change From Baseline in the Profile of Mood State (POMS) Scale at Week 12 Using LOCF
Description: The Profile of Mood States (POMS) Brief Form contains 30 adjectives; each participant is asked to rate the degree to which each adjective describes themselves based on how they felt during the past week including the date on which the adjective was rated. The possible ratings range from "0" (Not all all) to "4" (Extremely). The Total Mood Disturbance Score (range of 0 to 120) is obtained by summing the values of six domains. Higher scores indicate a more negative mood disturbance. The POMS was completed at Baseline (Day 1), and at the end of Weeks 4, 8, and 12 (or Early Termination).
Time Frame: Baseline to End of Treatment (Week 12)
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale | -7.3 (14.89) | -10.9 (17.97) | -11.5 (16.87)

21. Secondary Outcome: Change From Baseline in the Daytime Somnolence Score, an Item on the Medical Outcomes Study (MOS) Sleep Scale, at Week 12 Using LOCF
Description: The MOS Sleep Scale measures most constructs of sleep. The scale has a battery of questions to measure specific aspects of sleep in participants with co-morbidities. The four domains scored from the MOS Sleep Scale were "sleep disturbance,"' "sleep quantity,"' "sleep adequacy," and "daytime somnolence." The scores of the daytime somnolence domain ranged from 1 to 100, with a high score indicating greater daytime somnolence. The assessment was completed at Baseline (Day 1) and end of Weeks, 4, 8, and 12 (or end of Treatment).
Time Frame: Baseline and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 112 | 110
scores on a scale | -9.7 (20.39) | -9.8 (20.35) | -16.1 (19.58)

22. Secondary Outcome: Change From Baseline in the Sleep Disturbance Score, an Item on the MOS Sleep Scale, at Week 12 Using LOCF
Description: The MOS Sleep Scale measures most constructs of sleep. The scale has a battery of questions to measure specific aspects of sleep in participants with co-morbidities. The four domains scored from the MOS Sleep Scale were "sleep disturbance,"' "sleep quantity,"' "sleep adequacy," and "daytime somnolence." The scores of the sleep disturbance domain ranged from 1 to 100, with a high score indicating greater impairment of sleep. The assessment was completed at Baseline (Day 1) and end of Weeks, 4, 8, and 12 (or end of Treatment).
Time Frame: Baseline and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 112 | 110
scores on a scale | -17.0 (20.40) | -29.5 (23.27) | -30.7 (25.45)

23. Secondary Outcome: Change From Baseline in Sleep Adequacy, an Item on the MOS Sleep Scale, at Week 12 Using LOCF
Description: The MOS Sleep Scale measures most constructs of sleep. The scale has a battery of questions to measure specific aspects of sleep in participants with co-morbidities. The four domains scored from the MOS Sleep Scale were "sleep disturbance,"' "sleep quantity,"' "sleep adequacy," and "daytime somnolence." The scores of the sleep adequacy domain ranged from 1 to 100, with a high score indicating greater adequacy. The assessment was completed at Baseline (Day 1) and end of Weeks, 4, 8, and 12 (or end of Treatment).
Time Frame: Basline and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 112 | 110
scores on a scale | 13.6 (24.59) | 29.1 (29.91) | 27.7 (29.91)

24. Secondary Outcome: Change From Baseline in Sleep Quantity, an Item on the MOS Sleep Scale, at Week 12 Using LOCF
Description: The MOS Sleep Scale measures most constructs of sleep. The scale has a battery of questions to measure specific aspects of sleep in participants with co-morbidities. The four domains scored from the MOS Sleep Scale were "sleep disturbance,"' "sleep quantity,"' "sleep adequacy," and "daytime somnolence." The scores of the sleep quantity domain were measured in time (number of hours of sleep each night). The assessment was completed at Baseline (Day 1) and end of Weeks, 4, 8, and 12 (or end of Treatment).
Time Frame: Baseline and Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 111 | 110
hours | 0.3 (1.19) | 0.6 (1.25) | 0.8 (1.66)

25. Secondary Outcome: Change From Baseline in the Overall Life-Impact Score of the RLS Quality of Life (QoL) Questionnaire at Week 12 Using LOCF
Description: The Restless Legs Syndrome Quality of Life (RLS-QoL) questionnaire is a disease-specific, participant-rated questionnaire that assesses the impact of RLS on daily life, emotional well-being, social life, and work life of the participants. The RLS-QoL Questionnaire is presented on a 0 (lowest possible score) to 100 (highest possible score) scale. It was completed at Day 1 and at the end of Weeks 4, 8, and 12 (or Early Termination).
Time Frame: Baseline and Week 12
Population: MITT Population: The number of participants assessed varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
scores on a scale | 14.5 (15.74) | 19.3 (15.57) | 20.4 (17.14)

26. Secondary Outcome: Number of Participants Experiencing No RLS Symptoms in Each of the Seven 4-hour Periods From the 24-hour RLS Record at Week 12 (End of Treatment)
Description: RLS severity ratings were summarized in 6 non-overlapping 4-hour periods beginning at 8 AM. A 4-hour period from 6 PM to 10 PM was also prospectively included to reflect the time frame when the most participants would experience their first symptoms of the day.
Time Frame: Week 12
Population: MITT Population. The number analyzed represents participants within the MITT Population who reported no RLS symptoms at the end of Week 12.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 74 | 99 | 92
participants
  8 AM to 12 PM | 52 | 85 | 74
  12 PM to 4 PM | 51 | 74 | 69
  4 PM to 8 PM | 45 | 68 | 61
  6 PM to 10 PM | 39 | 55 | 55
  8 PM to 12 AM | 27 | 49 | 48
  12 AM to 4 AM | 38 | 74 | 67
  4 AM to 8 AM | 56 | 79 | 72

27. Secondary Outcome: Time to Onset of the First RLS Symptom From the 24-hour RLS Record Obtained at the End of Treatment (Week 12)
Description: The time to onset of the first RLS symptoms from the 24-hour RLS Record is defined as the length of time from the start of the 24-hour assessment period (8:00 AM) to the time when 50% of participants experienced their first symptom.
Time Frame: Week 12
Population: MITT Population. The number of participants assessed varies due to incomplete/missing data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Number analyzed (Participants) | 96 | 114 | 111
hours | 12.8 [9.5 to 15.0] | 13.5 [12.5 to 16.5] | 13.8 [11.5 to 17.0]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) and serious adverse event (SAE) collection started immediately following informed consent and continued throughout the study (up to Week 17).
Description: At the end of the follow-up period (30 days after the last day of taper [Day 119]), the study coordinator called participants (+/- 3 day window) who did not enroll in the open-label extension protocol to determine if any SAEs occurred, and the resolution date for any AEs that were ongoing at the end of the study.
Arm/Group | Placebo | GEn (XP13512/GSK1838262) 600 mg | GEn (XP13512/GSK1838262) 1200 mg
Serious Adverse Events (participants affected / at risk) | 1/96 | 2/115 | 0/111
Other Adverse Events (participants affected / at risk) | 36/96 | 68/115 | 64/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=96) | GEn (XP13512/GSK1838262) 600 mg (N=115) | GEn (XP13512/GSK1838262) 1200 mg (N=111)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Herniated Disc L5 (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=96) | GEn (XP13512/GSK1838262) 600 mg (N=115) | GEn (XP13512/GSK1838262) 1200 mg (N=111)
Somnolence (Nervous system disorders) | 2 | 25 | 20
Dizziness (Nervous system disorders) | 5 | 12 | 27
Headache (Nervous system disorders) | 8 | 17 | 15
Nasopharyngitis (Infections and infestations) | 7 | 13 | 11
Dry Mouth (Gastrointestinal disorders) | 2 | 5 | 9
Nausea (Gastrointestinal disorders) | 4 | 6 | 6
Fatigue (General disorders) | 5 | 6 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 9 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3
Sedation (Nervous system disorders) | 2 | 1 | 6
Sinus (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.